CLINICAL TRIAL: NCT05591755
Title: Evaluation of the Combination Drug Product Brimonidine Tartrate 0.025%/Ketotifen Fumarate 0.035% Ophthalmic Solution Compared to Its Components and Vehicle in an Allergen BioCube® in Subjects With Seasonal Allergic Conjunctivitis
Brief Title: Evaluation of Brimonidine Tartrate/Ketotifen Fumarate Combination in Adults With Seasonal Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 910
Record Dates: First submitted 2022-10-06; First posted 2022-10-24 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Seasonal Allergic Conjunctivitis
MeSH Terms: interventions — Brimonidine Tartrate; Ketotifen; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution (Experimental): Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution
  Interventions: Drug: Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution
- Ketotifen fumarate ophthalmic solution 0.035% (Experimental): Ketotifen fumarate ophthalmic solution 0.035%
  Interventions: Drug: Ketotifen fumarate ophthalmic solution 0.035%
- Brimonidine tartrate ophthalmic solution 0.025% (Experimental): Brimonidine tartrate ophthalmic solution 0.025%
  Interventions: Drug: Brimonidine tartrate ophthalmic solution 0.025%
- Vehicle ophthalmic solution (Experimental): Vehicle ophthalmic solution
  Interventions: Drug: Experimental: Vehicle ophthalmic solution

INTERVENTIONS:
Drug: Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution — Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution
  Arms: Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution
Drug: Ketotifen fumarate ophthalmic solution 0.035% — Ketotifen fumarate ophthalmic solution 0.035%
  Arms: Ketotifen fumarate ophthalmic solution 0.035%
Drug: Brimonidine tartrate ophthalmic solution 0.025% — Brimonidine tartrate ophthalmic solution 0.025%
  Arms: Brimonidine tartrate ophthalmic solution 0.025%
Drug: Experimental: Vehicle ophthalmic solution — Experimental: Vehicle ophthalmic solution
  Arms: Vehicle ophthalmic solution

SUMMARY:
To evaluate the efficacy of Combo compared to its individual components and compared to vehicle in a population of subjects with seasonal allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must:

  1. be at least 18 years of age of either sex and any race;
  2. provide written informed consent and sign the Health Information Portability and Accountability Act (HIPAA) form;
  3. be willing and able to follow all instructions and attend all study visits;
  4. provide proof of COVID-19 vaccination
  5. be able and willing to discontinue wearing contact lenses for at least 72 hours prior to Visit 2 and for the duration of the visit;
  6. have seasonal allergic conjunctivitis to ragweed or timothy grass documented by a self-reported history of ocular allergic symptoms for the last 2 consecutive years during the ragweed or timothy grass seasons and a positive skin test reaction to ragweed or timothy grass pollen as confirmed by the allergic skin test given at or within 24 months of the subject's Visit 1;
  7. (If female and of childbearing potential) agree to have urine pregnancy testing performed at visit 2, (must be negative); must not be lactating; and must agree to use at least 1 medically acceptable form of birth control throughout the study duration, for at least 14 days prior to and 1 month after receiving investigational drug. Acceptable forms of birth control are true abstinence (when this is in line with the preferred and usual lifestyle of the subject), spermicide with barrier, oral contraceptive, injectable or implantable method of contraception, transdermal contraceptive, intrauterine device, or surgical sterilization of male partner at least 3 months prior to receiving investigational drug (Visit 2). Note: Women considered capable of becoming pregnant include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy);
  8. (If male and with female partner of childbearing potential) must use at least 1 medically acceptable form of birth control· Note: Acceptable forms of birth control are true abstinence (when this is in line with the preferred and usual lifestyle of the subject) or vasectomy at least 3 months prior to receiving investigational drug (Visit 2). Without a vasectomy, must use condoms with spermicidal foam/gel/film/cream/suppository throughout the study duration, for at least 14 days prior to and 1 month after investigational drug (Visit 2).
  9. have a calculated visual acuity (VA) of 0.7 logMAR or better in each eye as measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart at Visit 1;
  10. have a positive Allergen BioCube challenge response to pollen exposure at the 90 minute time point of ABC exposure at Visit 2, defined as bilateral score of >2 in ocular itching and ocular redness.

Exclusion Criteria:

* Subjects may not:

  1. have known contraindications or sensitivities to the use of any of the investigational product medication or components;
  2. have a history of mild persistent, moderate or severe asthma within the preceding 5 years according to the National Heart, Blood, and Lung Institute classification (with the exception of exercise induced asthma).

     Note: Subjects with fall induced asthma that is either mild persistent (defined as >1 per week, but <1 per day), moderate persistent, or severe persistent will be excluded.
  3. have an upper respiratory tract or sinus infection within the previous 2 weeks of Visit 1;
  4. have a history of anaphylaxis or poor tolerability of previously administered allergen;
  5. have a compromised lung function at Visit 1 (defined as a peak expiratory flow rate [PEFR] that is below 80% of the predicted average PEFR, as calculated by gender, age, and measured height from the Mini-Wright instruction's table: Normal Adult Predicted Average Peak Expiratory Flow).
  6. have an abnormal blood pressure (defined as ≤ 90 or ≥ 160 (systolic) measured in mmHg or ≤ 60 or ≥ 100 (diastolic) measured in mmHg) at Visit 1;
  7. have any ocular condition that, in the opinion of the investigator, could affect the subject's safety or trial parameters (including but not limited to narrow angle glaucoma, clinically significant blepharitis, follicular conjunctivitis, iritis, pterygium, or a diagnosis of dry eye);
  8. have had ocular surgical intervention within three months prior to Visit 1, or during the trial or a history of refractive surgery six months prior to Visit 1, or have systemic surgery planned during the clinical trial or within 30 days after;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - 104 Butchertown Clinical Trials, Louisville, Kentucky
  - 101 Andover Eye Associates, Andover, Massachusetts
  - 105 - Advancing Vision Research, Goodlettsville, Tennessee
  - 102 Total Eye Care, PA, Memphis, Tennessee
  - 108 Emerson Clinical Research Institute Inc., Falls Church, Virginia
  - 107 Virginia Eye Institute, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each subject was randomized to receive one of the four treatments one time in both eyes
Groups:
- Vehicle Ophthalmic Solution: Experimental: Vehicle ophthalmic solution
Period: Overall Study
Arm/Group | Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution | Ketotifen Fumarate Ophthalmic Solution 0.035% | Brimonidine Tartrate Ophthalmic Solution 0.025% | Vehicle Ophthalmic Solution
Started | 58 | 57 | 58 | 56
Completed | 57 | 56 | 56 | 56
Not Completed | 1 | 1 | 2 | 0
Not completed — Screen Failure | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution (n = 56): Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution: Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution
- Ketotifen Fumarate Ophthalmic Solution 0.035% (n = 56): Ketotifen fumarate ophthalmic solution 0.035% (n = 56): Ketotifen fumarate ophthalmic solution 0.035% (n = 56)
- Brimonidine Tartrate Ophthalmic Solution 0.025% (n = 56): Brimonidine tartrate ophthalmic solution 0.025% (n = 56): Brimonidine tartrate ophthalmic solution 0.025% (n = 56)
- Vehicle Ophthalmic Solution (n = 56): Experimental: Vehicle ophthalmic solution (n = 56): Experimental: Vehicle ophthalmic solution (n = 56)
- Total: Total of all reporting groups
Arm/Group | Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution (n = 56) | Ketotifen Fumarate Ophthalmic Solution 0.035% (n = 56) | Brimonidine Tartrate Ophthalmic Solution 0.025% (n = 56) | Vehicle Ophthalmic Solution (n = 56) | Total
Number analyzed (Participants) | 57 | 56 | 58 | 56 | 227
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (15.06) | 35.0 (12.28) | 37.1 (16.05) | 37.1 (16.61) | 36.2 (15.03)
Age, Customized [Count of Participants; unit: Participants]
  Less than 65 years | 52 | 55 | 55 | 50 | 212
  Greater or equal to 65 years | 5 | 1 | 3 | 6 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 38 | 39 | 39 | 150
  Male | 23 | 18 | 19 | 17 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 14 | 14 | 15 | 55
  Not Hispanic or Latino | 45 | 42 | 44 | 41 | 172
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 10 | 12 | 10 | 44
  Asian | 1 | 3 | 1 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 9 | 12 | 35
  White | 36 | 36 | 34 | 31 | 137
  More than one race | 1 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 56 | 58 | 56 | 227

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching Symptom Score
Description: Ocular itching score evaluated by the subject at 10(±1), 30(±1), 60(±5), 360(±5), 420(±5), and 480(±5) minutes post-instillation of assigned IP at Visit 2 (0-4 scale, allowing half unit increments), with 4 is the worse outcome.
Time Frame: Assessed up to 480 minutes post-instillation of assigned IP
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution | Ketotifen Fumarate Ophthalmic Solution 0.035% | Brimonidine Tartrate Ophthalmic Solution 0.025% | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 57 | 56 | 58 | 56
score on a scale
  Visit 2, Before Qualification ABC | 0.175 (0.6031) | 0.085 (0.3136) | 0.267 (0.7549) | 0.098 (0.3493)
  Visit 2, 90 Minutes during Qualification ABC (Baseline) | 2.728 (0.5830) | 2.719 (0.5310) | 2.659 (0.4581) | 2.647 (0.5174)
  Visit 2, 10 min Post-Instillation | 1.807 (1.0501) | 1.808 (0.8712) | 1.991 (1.0163) | 2.022 (0.8302)
  Visit 2, 30 min Post-Instillation | 1.443 (0.8914) | 1.335 (0.8275) | 1.513 (1.0621) | 1.790 (0.8979)
  Visit 2, 60 min Post-Instillation | 1.110 (0.8737) | 1.205 (0.9171) | 1.220 (0.9425) | 1.438 (0.7720)
  Visit 2, 360 min Post-Instillation | 0.811 (0.8599) | 0.723 (0.7365) | 1.125 (0.9485) | 1.089 (1.0252)
  Visit 2, 420 min Post-Instillation | 0.851 (0.8568) | 0.656 (0.7348) | 1.078 (0.9461) | 0.978 (0.8624)
  Visit 2, 480 min Post-Instillation | 0.961 (1.0020) | 0.777 (0.8786) | 1.009 (0.9188) | 1.063 (0.9011)

2. Primary Outcome: Ocular Redness Measured by Ocular Itching Scale
Description: Ocular redness evaluated by the Investigator using slit lamp at 10(±1), 30(±1), 60(±5), 360(±5), 420(±5), and 480(±5) minutes post-instillation of assigned IP at Visit 2 (0-4 scale, allowing half unit increments), with 4 being the worse outcome.
Time Frame: Assessed up to 480 minutes post-instillation of assigned IP
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution | Ketotifen Fumarate Ophthalmic Solution 0.035% | Brimonidine Tartrate Ophthalmic Solution 0.025% | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 55 | 55 | 58 | 56
score on a scale
  Visit 2, Before Qualification ABC | 1.218 (0.5815) | 1.327 (0.5771) | 1.384 (0.5815) | 1.268 (0.6464)
  Visit 2, 90 Minutes during Qualification ABC (Baseline) | 2.469 (0.5430) | 2.500 (0.5045) | 2.642 (0.5832) | 2.478 (0.4984)
  Visit 2, 10 min Post-Instillation | 1.127 (0.8253) | 2.116 (0.6178) | 1.293 (0.8194) | 2.268 (0.6195)
  Visit 2, 30 min Post-Instillation | 0.934 (0.7388) | 1.911 (0.6421) | 1.103 (0.7609) | 2.165 (0.7011)
  Visit 2, 60 min Post-Instillation | 0.904 (0.6924) | 1.795 (0.7184) | 1.026 (0.7517) | 2.098 (0.6787)
  Visit 2, 360 min Post-Instillation | 1.316 (0.8245) | 1.723 (0.7608) | 1.405 (0.6896) | 1.955 (0.6416)
  Visit 2, 420 min Post-Instillation | 1.456 (0.7936) | 1.759 (0.7847) | 1.582 (0.6873) | 1.933 (0.6440)
  Visit 2, 480 min Post-Instillation | 1.553 (0.8125) | 1.929 (0.8471) | 1.832 (0.7757) | 2.063 (0.7043)

3. Secondary Outcome: Tearing Measured by Watery Eyes Scale
Description: Tearing evaluated by the subject at 10(±1), 30(±1), 60(±5), 360(±5), 420(±5), and 480(±5) minutes post-instillation of assigned IP at Visit 2 (0-4 scale, NOT allowing half unit increments), with 4 being the worse outcome.
Time Frame: up to 480 minutes post-instillation of assigned IP
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution | Ketotifen Fumarate Ophthalmic Solution 0.035% | Brimonidine Tartrate Ophthalmic Solution 0.025% | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 57 | 56 | 58 | 56
score on a scale
  Visit 2, Before Qualification ABC | 0.12 (0.503) | 0.04 (0.197) | 0.22 (0.773) | 0.13 (0.429)
  Visit 2, 90 Minutes during Qualification ABC (Baseline) | 1.34 (1.192) | 1.23 (0.977) | 1.41 (1.219) | 1.10 (0.997)
  Visit 2, 10 min Post-Instillation | 1.21 (1.056) | 1.10 (0.988) | 1.16 (1.056) | 1.14 (0.971)
  Visit 2, 10 min Post-Instillation change from baseline | -0.13 (0.961) | -0.13 (0.839) | -0.25 (0.768) | 0.04 (0.945)
  Visit 2, 30 min Post-Instillation | 0.77 (0.835) | 0.79 (0.883) | 0.94 (0.937) | 0.98 (0.958)
  Visit 2, 30 min Post-Instillation change from baseline | -0.57 (1.006) | -0.44 (0.826) | -0.47 (0.991) | -0.12 (0.853)
  Visit 2, 60 min Post-Instillation | 0.66 (0.757) | 0.65 (0.909) | 0.73 (0.865) | 0.76 (0.879)
  Visit 2, 60 min Post-Instillation change from baseline | -0.68 (0.989) | -0.58 (1.048) | -0.67 (1.024) | -0.34 (0.944)
  Visit 2, 360 min Post-Instillation | 0.42 (0.667) | 0.41 (0.668) | 0.64 (0.883) | 0.65 (0.744)
  Visit 2, 360 min Post-Instillation change from baseline | -0.92 (1.113) | -0.82 (0.811) | -0.77 (1.035) | -0.45 (1.030)
  Visit 2, 420 min Post-Instillation | 0.50 (0.726) | 0.34 (0.581) | 0.68 (0.945) | 0.46 (0.582)
  Visit 2, 420 min Post-Instillation change from baseline | -0.84 (1.123) | -0.89 (0.857) | -0.72 (1.085) | -0.64 (1.065)
  Visit 2, 480 min Post-Instillation | 0.54 (0.761) | 0.27 (0.539) | 0.56 (0.720) | 0.46 (0.785)
  Visit 2, 480 min Post-Instillation change from baseline | -0.81 (1.097) | -0.96 (0.830) | -0.84 (1.056) | -0.63 (1.102)

4. Secondary Outcome: Lid Swelling Measured by Eyelid Swelling Scale
Description: Lid swelling evaluated by the subject at 10(±1), 30(±1), 60(±5), 360(±5), 420(±5), and 480(±5) minutes post-instillation of assigned IP at Visit 2 (0-3 scale, NOT allowing half unit increments), with 3 being the worst outcome
Time Frame: up to 480 minutes post-instillation of assigned IP
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution | Ketotifen Fumarate Ophthalmic Solution 0.035% | Brimonidine Tartrate Ophthalmic Solution 0.025% | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 57 | 56 | 58 | 56
score on a scale
  Visit 2, Before Qualification ABC | 0.09 (0.434) | 0.00 (0.000) | 0.11 (0.409) | 0.04 (0.187)
  Visit 2, 90 Minutes during Qualification ABC (Baseline) | 1.04 (0.972) | 0.70 (0.883) | 1.05 (0.921) | 0.92 (0.873)
  Visit 2, 10 min Post-Instillation | 0.85 (0.973) | 0.77 (0.874) | 1.03 (0.957) | 0.98 (0.904)
  Visit 2, 10 min Post-Instillation change from baseline | -0.18 (0.748) | 0.07 (0.606) | -0.03 (0.652) | 0.06 (0.714)
  Visit 2, 30 min Post-Instillation | 0.75 (0.851) | 0.75 (0.905) | 0.72 (0.750) | 0.90 (0.881)
  Visit 2, 30 min Post-Instillation change from baseline | -0.28 (0.851) | 0.05 (0.644) | -0.34 (0.740) | -0.02 (0.798)
  Visit 2, 60 min Post-Instillation | 0.65 (0.802) | 0.64 (0.841) | 0.59 (0.744) | 0.81 (0.902)
  Visit 2, 60 min Post-Instillation change from baseline | -0.39 (0.835) | -0.05 (0.644) | -0.47 (0.805) | -0.11 (0.785)
  Visit 2, 360 min Post-Instillation | 0.48 (0.762) | 0.43 (0.817) | 0.61 (0.864) | 0.67 (0.886)
  Visit 2, 360 min Post-Instillation change from baseline | -0.55 (0.817) | -0.27 (0.707) | -0.44 (0.869) | -0.25 (0.929)
  Visit 2, 420 min Post-Instillation | 0.60 (0.832) | 0.44 (0.695) | 0.61 (0.838) | 0.61 (0.824)
  Visit 2, 420 min Post-Instillation change from baseline | -0.44 (0.921) | -0.26 (0.681) | -0.44 (0.822) | -0.31 (0.877)
  Visit 2, 480 min Post-Instillation | 0.55 (0.777) | 0.42 (0.731) | 0.55 (0.826) | 0.58 (0.857)
  Visit 2, 480 min Post-Instillation change from baseline | -0.48 (0.802) | -0.28 (0.750) | -0.50 (0.827) | -0.34 (0.895)

5. Secondary Outcome: Chemosis Evaluated
Description: Chemosis evaluated by the Investigator using slit lamp at 10(±1), 30(±1), 60(±5), 360(±5), 420(±5), and 480(±5) minutes post-instillation of assigned IP at Visit 2 (0-4 scale, allowing half unit increments), with 4 being the worse outcome.
Time Frame: up to 480 minutes post-instillation of assigned IP
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution | Ketotifen Fumarate Ophthalmic Solution 0.035% | Brimonidine Tartrate Ophthalmic Solution 0.025% | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 57 | 56 | 58 | 56
score on a scale
  Visit 2, Before Qualification ABC | 0.000 (0.0000) | 0.000 (0.0000) | 0.004 (0.0328) | 0.022 (0.1372)
  Visit 2, 90 Minutes during Qualification ABC (Baseline) | 0.298 (0.7249) | 0.143 (0.3626) | 0.134 (0.3811) | 0.129 (0.3843)
  Visit 2, 10 min Post-Instillation | 0.228 (0.5830) | 0.121 (0.3371) | 0.086 (0.2502) | 0.156 (0.4537)
  Visit 2, 10 min Post-Instillation change from baseline | -0.070 (0.3196) | -0.022 (0.2490) | -0.047 (0.1957) | 0.027 (0.3804)
  Visit 2, 30 min Post-Instillation | 0.158 (0.5274) | 0.094 (0.3110) | 0.039 (0.1609) | 0.134 (0.4290)
  Visit 2, 30 min Post-Instillation change from baseline | -0.140 (0.4092) | -0.049 (0.2877) | -0.095 (0.2683) | 0.004 (0.5319)
  Visit 2, 60 min Post-Instillation | 0.154 (0.5298) | 0.094 (0.2883) | 0.052 (0.1973) | 0.112 (0.3597)
  Visit 2, 60 min Post-Instillation change from baseline | -0.145 (0.4405) | -0.049 (0.2450) | -0.082 (0.2406) | -0.018 (0.4764)
  Visit 2, 360 min Post-Instillation | 0.114 (0.3662) | 0.094 (0.2960) | 0.069 (0.2556) | 0.089 (0.2756)
  Visit 2, 360 min Post-Instillation change from baseline | -0.184 (0.5561) | -0.049 (0.3706) | -0.065 (0.2321) | -0.040 (0.4258)
  Visit 2, 420 min Post-Instillation | 0.105 (0.3502) | 0.067 (0.2050) | 0.082 (0.2624) | 0.076 (0.2608)
  Visit 2, 420 min Post-Instillation change from baseline | -0.193 (0.5408) | -0.076 (0.2564) | -0.052 (0.2555) | -0.054 (0.4439)
  Visit 2, 480 min Post-Instillation | 0.088 (0.3006) | 0.076 (0.2232) | 0.091 (0.2678) | 0.058 (0.2184)
  Visit 2, 480 min Post-Instillation change from baseline | -0.211 (0.5505) | -0.067 (0.2919) | -0.043 (0.2815) | -0.071 (0.4490)

ADVERSE EVENTS:
Time Frame: Assessed for approximately 8 hours after treatment
Description: Ocular Adverse events were reported at the participant level
Arm/Group | Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution | Ketotifen Fumarate Ophthalmic Solution 0.035% | Brimonidine Tartrate Ophthalmic Solution 0.025% | Vehicle Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/56 | 0/58 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/56 | 0/58 | 0/56
Other Adverse Events (participants affected / at risk) | 1/57 | 6/56 | 2/58 | 5/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brimonidine Tartrate 0.025%/ Ketotifen Fumarate 0.035% Ophthalmic Solution (N=57) | Ketotifen Fumarate Ophthalmic Solution 0.035% (N=56) | Brimonidine Tartrate Ophthalmic Solution 0.025% (N=58) | Vehicle Ophthalmic Solution (N=56)
Visual acuity reduced (Eye disorders) | 1 | 2 | 2 | 2
Ocular hyperaemia (Eye disorders) | 0 | 2 | 0 | 1
Eyelid exfoliation (Eye disorders) | 0 | 0 | 0 | 1
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 1
Conjunctival oedema (Eye disorders) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT05591755/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/55/NCT05591755/SAP_001.pdf